CLINICAL TRIAL: NCT00852059
Title: Effect of Methylphenidate Formulation on ADHD-patients' Adherence to Medical Treatment. A Comparison of Medikinet Retard® (ER) Once Daily and Medikinet® (IR) Twice Daily in Children and Adolescents Diagnosed With ADHD
Brief Title: Adherence to Stimulant Treatment in Attention-Deficit Hyperactivity Disorder (ADHD) Patients (ASTA)
Acronym: ASTA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Diffculties to recruit anticipated study size, now analysis
Sponsor: Prof. Huss (Other)
Responsible Party: Sponsor-Investigator, Prof. Huss, Prof. Dr. Michael Huss, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JoGu_KJP_ASTA-3285-26
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: ADHD
Keywords: ADHD; children; adolescents; methylphenidate; adherence; immediate release; extended release; efficacy
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate release (Experimental): Treatment with immediate release (IR) methylphenidate (Medikinet®) in the morning and 3-4 h later (twice a day)
  Interventions: Drug: Immediate release methylphenidate (Medikinet®)
- Extended release (Active Comparator): Treatment with extended release (ER) methylphenidate (Medikinet reatard®) applied with breakfast(once daily)
  Interventions: Drug: Extended release methylphenidate (Medikinet retard®)

INTERVENTIONS:
Drug: Immediate release methylphenidate (Medikinet®) — Treatment: methylphenidate in the morning and 3-4 h later (twice daily), immediate release
  Other Names: Medikinet®
  Arms: Immediate release
Drug: Extended release methylphenidate (Medikinet retard®) — Treatment: methylphenidate applied with breakfast(once daily), extended release
  Other Names: Medikinet retard®
  Arms: Extended release

SUMMARY:
This study determined to measure non-adherence assessed by the number of non-adherent days during the clinical trial of 100 days using the Medication Event Monitoring System (MEMS).

Study Design:

* prospective
* multi-centric
* open-label
* randomized
* active-controlled trial

DETAILED DESCRIPTION:
The study is designed as a prospective, multi-centric, open-label, randomized, active-controlled trial. ADHD-children and adolescents of both sexes, 6-17 of age, effectively treated with stimulants are recruited in two centres. Over a naturalistic run-in phase of four weeks adherence to medication taken before randomisation is measured. In the subsequent controlled clinical trial 50% of the participants are randomized to extended release (ER) methylphenidate (Medikinet retard®) applied with breakfast, 50% are randomized to immediate release (IR) methylphenidate (Medikinet®) in the morning and 3-4 h later (clinical trial). To optimize ecological validity, no double-dummy technique is applied; the allocation to either study arm is non-blinded.

According to the power calculation 106 patients will be randomized. The total duration of the study is 18 months. Starting with a run-in visit, each eligible patient is observed in the naturalistic run-in phase for four weeks. Subsequently, patients participate 100 days in the clinical trial starting with a baseline visit, an in between-visit and a final visit. Medical care is provided in the routine program of both study centres. To record the adherence, medication events are counted by Medication Event Monitoring System (MEMS).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (separately for children aged 6-11 years and 12-17 years)
* Children and adolescents of both sexes aged 6 - 17 years
* Confirmed diagnosis of ADHD by semi structured-clinical interview K-SADS
* ADHDRS-IV-Parent Version (18-Item-Scale) raw score ≥ 1,5 SD above norm under non-medicated conditions (either drug holiday or prior to medication within the past 6 months)
* Effective treatment with a stable dose of methylphenidate for at least one month (max. 60 mg/day) proved by a 25% symptom reduction in ADHD-RS under medication, compared to retrospective ADHD-RS without medication within the past 6 months.
* Acceptance and capability to swallow capsules of product size, proved by an equally sized placebo provided by Medice®.
* Sufficient knowledge of the German language
* Adequate contraception in case of sexual activity

Exclusion Criteria:

* Contraindications against methylphenidate
* Previous stable methylphenidate intake more than twice daily
* All severe psychiatric disorders except oppositional defiant disorder (ODD) or conduct disorder. In order to reflect the usual co-morbid spectrum of ADHD, mild or moderate anxiety or depressive disorders are accepted in the study.
* All severe somatic diseases as assessed by the baseline examination or medical history (including life-time history of epileptic disorders)
* Pathological results for vital signs, blood pressure and pulse
* Reported pathological results for ECG during the last 12 months
* Reported pathological results for differential blood count and hepatic metabolism during the last 6 months
* Indication for hospitalization
* Suicidality (assessed by MADRS Item 10, Score ≥ 3)
* IQ < 70 (clinically assessed)
* Any psychotropic co-medication
* Detention in an institution on official or judicial ruling
* Unwillingness to transmit pseudonym data according to German regulations
* Simultaneous participation in another clinical trial according to German Drug Law (AMG)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Non-adherence assessed by the number of non-adherent days during the clinical trial of 100 days using the Medication Event Monitoring System (MEMS) | 100 days

SECONDARY OUTCOMES:
Number of non-adherent days measured by pill count | 100 days
Time interval until a total number of 30 days of non-adherence is reached cumulatively during the clinical trial measured by MEMS | 100 days
Quality of life during measured by Child Health Illness Profile - Child Edition (CHIP-CE) Score | 100 days
The efficacy of stimulant treatment during the clinical trial measured by ADHD-Rating Scale- Parent Version Sum Score | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Huss, Prof. Dr., Principal Investigator — Johannes Gutenberg University, Mainz, Dep. of Child and Adolescent Psychiatry
Locations (1):
- Universitätsmedizin der Johannes Gutenberg-Universität Mainz - Körperschaft des öffentlichen Rechts, Mainz, Germany